CLINICAL TRIAL: NCT01506024
Title: Minimal Invasive Surgery in Total Hip Arthroplasty Patients; Short- and Long Term Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/450
Record Dates: First submitted 2011-12-09; First posted 2012-01-09 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Hip Osteoarthritis
Keywords: Arthroplasty, Replacement, Hip; Surgical Procedures, Operative; Surgical Procedures, Minimally Invasive
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip; Tacrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THA Direct lateral (Active Comparator): Total hip arthroplasty (THA) carried out by direct lateral approach (DLA)
  Interventions: Procedure: Total hip arthroplasty direct lateral approach
- THA Posterior (Experimental): Total hip arthroplasty (THA) carried out by posterior approach (DLA)
  Interventions: Procedure: Total hip arthroplasty posterior approach
- THA Anterior (Experimental): Total hip arthroplasty (THA) carried out by anterior approach (DLA)
  Interventions: Procedure: Total hip arthroplasty, anterior approach

INTERVENTIONS:
Procedure: Total hip arthroplasty direct lateral approach
  Other Names: Total hip replacement; THA
  Arms: THA Direct lateral
Procedure: Total hip arthroplasty posterior approach
  Other Names: Total hip replacement; THA
  Arms: THA Posterior
Procedure: Total hip arthroplasty, anterior approach
  Other Names: Total hip replacement; THA
  Arms: THA Anterior

SUMMARY:
The aim of the present study is to explore the most efficient surgical approach in total hip replacement in short and long term when concerning strength, functionality and postoperative complications.

The objective is to register muscular strength, hip joint functionality/mobilisation and complications after total hip arthroplasty (THA) performed by the direct lateral approach (DLA), the posterior approach (PA) and the anterior approach (AA). The latter is a modified Smith-Petersen approach which follows the principles of minimally invasive surgery (MIS).

The primary working hypothesis is that due to a minimal dissection and reduced trauma in the muscles, patients will tolerate early hospital discharge better after the AA than the PA and the DLA. Patients in the AA group are also thought to be more active and maintain muscular strength and hip joint functionality/mobilisation better than patients in the lateral group.

DETAILED DESCRIPTION:
With total hip replacement surgery, the orthopaedic surgeon's aim is not only pain relief for the patient, but also restoration of hip joint biomechanics resulting in a minimal functional deficit and maximal longevity of the implant. It is not exceptional that these patients still experience mild to moderate long-term impairments postoperatively. These impairments include pain, muscle weakness of the hip abductors, contracture of the hip, gait disorders, as well as weakness of hip extensors and flexors. These problems may in turn lead to complications such as joint instability and loosening of the implant.

MIS is defined as a surgical approach performed through a short skin and muscle incision to avoid injury to muscles and tendons. Following minimally invasive approach reduced muscle trauma has been found. Moreover clinical outcome improved, as the gluteus medius muscle can be spared more successfully. However, it is debated whether or not the overall results of MIS are superior, or even as good as the traditional hip replacement surgery in terms of component placing and time to revision of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for THA
* Diagnosis of primary osteoarthritis as the main cause for elective THA
* American Society of Anesthesiologists (ASA) score I, II, and stable III

Exclusion Criteria:

* Musculoskeletal diseases
* Current heart/pulmonary- or malignant diseases likely to influence the physical testing performance.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 3 months postoperatively
  Measured by 1 repetition maximum (1 RM)

SECONDARY OUTCOMES:
Hip joint functionality and mobility | 3 months postoperatively
  Measured by patient completed questionnaires and clinician reported scores
activity level | 6 subsequent days postoperatively
  Measured by an activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Winther SB, Husby VS, Foss OA, Wik TS, Svenningsen S, Engdal M, Haugan K, Husby OS. Muscular strength after total hip arthroplasty. A prospective comparison of 3 surgical approaches. Acta Orthop. 2016 Feb;87(1):22-8. doi: 10.3109/17453674.2015.1068032. Epub 2015 Aug 27. PMID 26141371
- [Result] Winther SB, Foss OA, Husby OS, Wik TS, Klaksvik J, Husby VS. Muscular strength and function after total hip arthroplasty performed with three different surgical approaches: one-year follow-up study. Hip Int. 2019 Jul;29(4):405-411. doi: 10.1177/1120700018810673. Epub 2018 Nov 13. PMID 30421633